CLINICAL TRIAL: NCT07171866
Title: From Esthetics to Function: Can Socket Shield Technique Prove Long-term Effectiveness Either With Immediate or Delayed Implant Placement Protocols? A 6-Year Randomized Clinical Trial
Brief Title: Socket Shield Technique for Immediate and Delayed Implant Placement: A 6-Year Clinical Tria
Acronym: SST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, Lecturer of Oral and Maxillofacial Surgery, Faculty of Dentistry, Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.25.09.21
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Ridge Preservation; Implant Dentistry
Keywords: Socket Shield Technique; Immediate Implant Placement; Delayed Implant Placement; CBCT; Ridge Width Change; Pink Esthetic Score; Alveolar Ridge Preservation; Long-term Implant Outcomes

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel groups: one receiving immediate implant placement and the other delayed placement following the SST. Each group followed the assigned intervention protocol throughout the study.
Who Masked: Outcomes Assessor
Masking Description: The radiographic outcomes assessor was blinded to group allocation. No other masking was implemented due to the surgical nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Implant Placement with SST (Active Comparator): Participants received the SST with immediate implant placement performed at the time of extraction.
  Interventions: Procedure: Immediate Implant Placement with SST
- Delayed Implant Placement with SST (Active Comparator): Participants received the SST with delayed implant placement, performed 6 months after extraction and shield preparation.
  Interventions: Procedure: Delayed Implant Placement with SST

INTERVENTIONS:
Procedure: Immediate Implant Placement with SST — Participants underwent extraction and socket shield preparation, followed by immediate implant placement in the esthetic maxillary zone. The implant was inserted at the same surgical session using a flapless or minimally invasive approach. CBCT was used to guide planning and assess ridge dimensions. Healing and follow-up assessments were conducted at 1 year and 6 years post-placement.
  Arms: Immediate Implant Placement with SST
Procedure: Delayed Implant Placement with SST — Participants underwent extraction and socket shield preparation. Implant placement was delayed for 6 months to allow soft and hard tissue healing. The implant was placed after verifying shield stability and ridge preservation via CBCT. Follow-up assessments were conducted at 1 year and 6 years post-placement.
  Arms: Delayed Implant Placement with SST

SUMMARY:
This study investigates the long-term performance of the Socket Shield Technique (SST) for preserving the bone and soft tissue around dental implants when used with two different timing protocols: immediate versus delayed implant placement.

SST is a surgical technique where a thin portion of the tooth root (the buccal shield) is intentionally retained to support the facial bone and gum tissues after tooth extraction. While SST is known to enhance esthetics and preserve bone in the short term, little evidence exists on its long-term effectiveness in different clinical scenarios.

This randomized clinical trial enrolled patients who needed single-tooth implants in the esthetic zone. Participants were randomly assigned to one of two groups:

Immediate SST group: the implant was placed at the same time the socket shield was prepared.

Delayed SST group: implant placement was performed six months after socket shield preparation.

Over a 6-year follow-up period, both groups were evaluated for:

Changes in ridge width and bone height using CBCT imaging. Esthetic outcomes using the Pink Esthetic Score (PES). Patient satisfaction through a structured questionnaire.

The goal is to determine whether SST offers reliable long-term outcomes in either immediate or delayed implant placement scenarios, supporting its broader clinical use.

DETAILED DESCRIPTION:
This randomized controlled clinical trial was conducted to compare the long-term clinical, radiographic, esthetic, and patient-reported outcomes of the SST when used with either immediate or delayed implant placement in the anterior maxilla.

Study Design:

Parallel-arm, randomized controlled trial Conducted at the Faculty of Dentistry, Mansoura University Sample: 25 patients needing single-tooth replacement

Groups:

Immediate SST: implant placed at time of shield preparation Delayed SST: implant placed after 6-month healing

Primary Outcome:

Ridge Width Change: measured at 1 mm, 2 mm, 4 mm, and 6 mm apical to the implant platform using standardized CBCT imaging at baseline, 1 year, and 6 years.

Secondary Outcomes:

Buccal/Palatal Bone Height Implant Stability Pink Esthetic Score Patient Satisfaction

Serial CBCT scans were superimposed using the Fusion module of OnDemand3D software for precise assessment. All clinical assessments were performed by calibrated, blinded examiners. Statistical analysis was performed using SPSS, with significance set at p < 0.05.

This study provides one of the first long-term comparative evaluations of SST in different implant placement protocols, offering evidence to support its clinical reliability over a 6-year period.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring single-tooth replacement in the anterior maxilla (esthetic zone)
* Age between 18-65 years
* Good systemic health
* Demonstrated good oral hygiene
* Presence of an intact buccal plate
* Class I or II sagittal root position
* Sufficient apical bone volume and quality for implant placement
* Willingness and ability to comply with study protocol and follow-up schedule
* Signed informed consent

Exclusion Criteria:

* Presence of acute infection at the extraction site (e.g., abscess)
* Vertical root fracture or advanced periodontitis with buccal plate loss
* Uncontrolled systemic disease (e.g., diabetes, osteoporosis)
* Parafunctional habits (e.g., bruxism, clenching)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Horizontal Ridge Width Change at 1, 2, 4, and 6 mm Apical to the Implant Platform | Immediately after implant placement (baseline), 1 year, and 6 years post-placement
  Ridge width was measured at 1 mm, 2 mm, 4 mm, and 6 mm apical to the implant platform using standardized CBCT scans. Superimposed scans were aligned using the Fusion module of OnDemand3D™ software. Changes in horizontal ridge width were calculated by subtracting baseline values from those at 1 year and 6 years to assess dimensional stability over time.
  Unit of Measure: → Millimeters (mm) Safety Issue: → No

SECONDARY OUTCOMES:
Buccal and Palatal Bone Height Change | Immediately after implant placement (baseline), 1 year, and 6 years post-placement
  Bone height was measured from the implant apex to the most coronal point of the buccal and palatal bone crest using CBCT. Changes were calculated at each follow-up relative to baseline.
  Unit of Measure: → Millimeters (mm) Safety Issue: → No
Implant Stability Quotient (ISQ) | Immediately after implant placement, loading time and 1-year post-placement
  Implant stability was assessed using a resonance frequency analysis device (Osstell ISQ). Buccolingual and mesiodistal values were averaged to calculate ISQ.
  Unit of Measure:
  → ISQ Units
  Safety Issue:
  → No
Pink Esthetic Score (PES) | At implant loading, 1 year, and 6 years post-placement
  The esthetic outcome was assessed using the PES, evaluating five parameters each scored from 0-2. Total PES ranges from 0-10, with ≥6 considered clinically acceptable.
  Unit of Measure: → Score (0-10) Safety Issue: → No
Patient Satisfaction (VAS Score) | At implant loading, 1 year, and 6 years post-placement
  Satisfaction was measured using a 100 mm visual analog scale (VAS) on three dimensions: overall experience, expectations, and esthetics. Scores were converted into percentages.
  Unit of Measure: → VAS (%) Safety Issue: → No

CONTACTS AND LOCATIONS:
Overall Officials: Soaad Tolba Badawy, Lecturer, Oral Surgery, MU, Principal Investigator — Faculty of dentistry, Mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to privacy considerations, and limitations in participant consent regarding external data sharing.